CLINICAL TRIAL: NCT04667806
Title: Study of the Quality of Life in Surviving Lung Transplant Patients Between 2008 and 2018 by SF36 and St Georges's Questionnaires
Brief Title: Health Related Quality of Life in Lung Transplantation in Strasbourg
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7952
Record Dates: First submitted 2020-11-24; First posted 2020-12-16 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Lung Transplantation
Keywords: Health related quality of life; Lung transplantation; SF36; St Georges's Respiratory
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Questionnaires — Use questionnaires ( SF36 questionnaire (generic score) and St Georges's questionnaire (specific score))

SUMMARY:
The aim of this study is to study the quality of life in lung transplant patients. The cohort includes all of the surviving and transplanted patients at the New Civil Hospital in Strasbourg between 2008 and 2018. The main objective is to assess the quality of life of this cohort by two questionnaires which are the SF36 (generic score) and the saint Georges's questionnaire (specific score).

The secondary objectives are the measurement of survival after lung transplantation, the comparison of the quality of life of these patients with that of the general population by the SF36 questionnaire, the search for perioperative factors influencing the quality of life and finally the search for an association between quality of life and socio-professional life.

ELIGIBILITY:
Inclusion Criteria:

* Transplants survivors in Strasbourg hospital between 2008 et 2018
* Patient able to answer a questionnaire in french

Exclusion Criteria:

* Pregnancy
* Vulnerability
* Safeguard of justice, curatorship or tutorship
* Emergency situation
* Difficilty in understanding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Transplants survivors in Strasbourg hospital between 2008 et 2018
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life | 12 month
  Score obtained by a questionnaire : SF36
Health related quality of life | 12 month
  Score obtained by a questionnaire : St Georges

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided